CLINICAL TRIAL: NCT04505709
Title: STOP-Coronavirus: Clinical, Immunological, Genomic, Virological and Bioethical Actors of COVID-19
Brief Title: Clinical, Immunological, Genomic, Virological and Bioethical Actors of COVID-19
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Collaborators: Hospital Universitario 12 de Octubre (Other); Fundacion Investigacion Biomedica Hospital 12 de Octubre (Unknown); Hospital Universitario Fundación Jiménez Díaz (Other); Hospital Universitario Infanta Elena (Unknown); Hospital Universitario Virgen de la Arrixaca (Other); Instituto Murciano de Investigación Biosanitaria Virgen de la Arrixaca (Other)
Responsible Party: Sponsor
Other Study IDs: STOP-Coronavirus; COV20/00181 (Other Grant/Funding Number: Instituto de Salud Carlos III)
Record Dates: First submitted 2020-08-07; First posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Covid19
Keywords: genomics; bioethics; SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — SARS-CoV-2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The STOP-Coronavirus project is an integrated and multidisciplinary study that aims to analyze the impact that various factors have on the evolution and prognosis of the current COVID-19. Clinical presentation, immunological markers, therapeutic strategies, host and virus genomics, and bioethical considerations will be analyzed with a prospective multicenter cohort of patients with a diagnosis of COVID-19.

DETAILED DESCRIPTION:
This project led my Dr Aguado Garcia, has established 8 Work Parckages (WP) to analyze factors involved in the impact of COVID-19. WP that correspond to University Hospital Fundacion Jimenez Diaz are described in this register across different objectives:

WP 3 (Dr Ayuso García) is aimed to analyze the genetic markers of host susceptibility associated with clinical evolution of COVID-19.

WP 6 (Dr Ruiz Hornillos) will study the socio-economic and bioethical repercussions of COVID-19.

WP 7 (Dr Perales) will analyze the complexity of the spectrum of SARS-CoV-2 mutants and their possible association with the evolutionary course of COVID-19

This project will guide and individualize the clinical and therapeutic approach to COVID-19 and mitigate the health and social impact of the pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of COVID-19 (positive RT-PCR for SARS-CoV-2 in respiratory sample).

Exclusion Criteria:

* Suspected coronavirus infection without diagnostic confirmation

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with confirmed diagnosis of COVID-19 (positive RT-PCR for SARS-CoV-2 in respiratory sample) will from the following university hospitals, will be enrolled for the study:
  Hospital Universitario 12 de Octubre, Hospital Universitario Fundación Jiménez Díaz, Hospital Universitario Infanta Elena, Hospital Clínico Universtario Virgen de la Arrixaca
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Identification of host genetic markers associated with the evolution of COVID-19 | 4 months
  Based on the cohort of patients with a confirmed diagnosis of COVID-19 and according to severity categories, a Genome-wide association study (GWAS) will be carried out
Analysis of bioethical aspects related to in-hospital management of the health crisis | 10 months
  Through structured interviews, data collection in each epidemiological period, and evaluation of the application of recommended measures from the bioethical point of view, a comparative study will be carried out between hospitals, taking into account the use of resources and analyzing the situations of ethical commitment for healthcare professionals, patients and institutions
Analysis of the spectrum of mutants of SARS-CoV-2 and its possible association with the clinical evolution of COVID-19 | 6 months
  From the mass sequencing of SARS-CoV-2 and the calculation of viral variability indices, it will be studied whether or not there is an association between the spectrum of viral mutants and clinical evolution

CONTACTS AND LOCATIONS:
Locations (1):
- Fundacion Jimenez Diaz, Madrid, Spain